CLINICAL TRIAL: NCT04168216
Title: A 12-week Exploratory Study to Characterise the RelatiOnship Between Changes in InflammatoRy Markers, Lung Function, Symptoms And ReLiever Use in Chronic Obstructive Pulmonary Disease Patients (CORAL)
Brief Title: Study of Relationship Between Changes in Inflammation, Lung Function, Symptoms and Medication Use in COPD Patients
Acronym: CORAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: D6930R00002
Record Dates: First submitted 2019-10-11; First posted 2019-11-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, sputum, nasal and urine samples will be collected for exploratory research.
  Blood samples will be collected for future genetic/DNA research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intention with the study is to have a better understanding of what happens to COPD patients' symptoms, lung function and markers of inflammation over 12 weeks. This information will increase the understanding of COPD and how to design new treatments for COPD in the future.

DETAILED DESCRIPTION:
This is a Phase IV, open-label, single-arm, single-site study. The purpose of this exploratory study is to gain longitudinal insights into the relationships between the inflammatory profile, symptoms, lung function, and reliever use in subjects with chronic obstructive pulmonary disease (COPD).

The study will include a minimum of 8 clinic visits and consist of a Screening Visit (Visit 1), a 4-week run-in period, a Baseline Visit (Visit 2) and a 12-week observational period, including 6 visits scheduled every 2 weeks. To standardise the use of COPD medications all subjects will receive maintenance Duaklir and reliever Ventolin for the duration of the study. During the observational period, additional visits may occur if subjects experience a worsening of their COPD symptoms. For each individual subject, the duration of participation in the study will be 16 weeks.

Estimated study duration is approximately 20 months including approximately 50 patients.

ELIGIBILITY:
Inclusion Criteria for Entry in the Run-in Period:

1. Provision of signed and dated, written ICF prior to any study specific procedures, sampling, and analyses (at Visit 1).
2. Male or female subjects ≥40 years of age at the time of signing the ICF.
3. A physician diagnosis of COPD and receiving maintenance treatment with a LABA in combination with an ICS, a LAMA, or both (ie, LABA+ICS, LABA+LAMA, or LABA+ICS+LAMA), for at least 3 months prior to Visit 1.
4. Physician-documented prescription and subject-confirmed use of an inhaled short-acting bronchodilator (β2 agonists or anticholinergics) as rescue medication prior to study.
5. Current or ex-smoker with ≥10 pack-year history.
6. Post-bronchodilator FEV1/FVC <0.7 recorded in medical history.
7. Blood eosinophils >0.1×109 cells/L.
8. The subject must be able to read, speak, and understand English; and be able to, in the Investigator's judgment, comply with the Study Protocol.
9. Negative pregnancy test (urine) for female subjects of childbearing potential at Visit 1

Incusion Criteria for Entry in the Observational Period:

1. Frequent use of SABA (≥200 µg of Ventolin per day, for at least 75% of days in the 3 weeks prior to Visit 2).
2. At least 70% compliance with daily FeNO, spirometry, EXACT, and BCSS during the last 3 weeks prior to Visit 2.
3. Blood eosinophils >0.1×109 cells/L at Visit 2.
4. Negative pregnancy test (urine) for female subjects of childbearing potential at Visit 2.

Exclusion Criteria:

1. As judged by the Investigator, any evidence of drug/substance abuse which would pose a risk to subject safety, interfere with the conduct of study, have an impact on the study results, or affect the subject's ability to participate in the study.
2. Concurrent Respiratory Disease: Presence of a known pre-existing, clinically important lung condition other than COPD.
3. Concurrent diagnosis of asthma (subjects with a history of asthma may be included).
4. Any disease currently treated with chronic oral/systemic corticosteroids.
5. Subjects with a history/treatment of malignancy, and which in the Investigator's opinion could compromise the safety of the subject.
6. Other Concurrent Medical Conditions: Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
7. Subjects currently treated with eosinophil-depleting medications (ie, mepolizumab, benralizumab), or who have been treated within 5.5 half-lives of eosinophil-depleting medications.
8. Subjects who have had a COPD exacerbation requiring oral corticosteroids and/or antibiotics in the last 30 days before the run-in period. Subjects will be able to be re-screened 30 days following an exacerbation.
9. Participation in another clinical study with any marketed or investigational biologic drug within 4 months or 5 half-lives (whichever is longer) prior to Visit 1.
10. Participation in another clinical study with a non-biologic investigational product or new formulation of a marketed non-biologic drug during the last 30 days prior to Visit 1 that, in the opinion of the Investigator, could impact the results of the current study.
11. Subjects with a known hypersensitivity to the treatment or any of the excipients of Duaklir and Ventolin.
12. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
13. Judgment by the Investigator that the subject should not participate in the study if the subject is unlikely to complete the observational period (eg, literacy, substance abuse, life-threatening comorbidity).
14. Previous entry into the observation period in the present study.
15. For women only - currently pregnant (confirmed with positive pregnancy test), breast-feeding or planned pregnancy during the study. Women of childbearing potential not using acceptable contraceptive measures, as judged by the Investigator.
16. As judged by the Investigator, planned hospitalisation/vacation during the study that interferes with study assessments.

    -

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients diagnosed with symptomatic COPD and blood eosinophil count >0.1×109 cells/L, who are receiving maintenance treatment with a long-acting β2 agonist (LABA) in combination with ICS and/or a long-acting muscarinic antagonist (LAMA) and require use of an inhaled short-acting bronchodilator (β2 agonists or anticholinergics) as rescue medication. The study will include both current and former smokers (with at least 10 pack-year history) and intends to recruit a maximum of 30% current smokers.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Inflammation data will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Inflammation:
  FeNO (daily) Blood eosinophils, CRP, and EDN (fortnightly) Sputum eosinophils and neutrophils (weekly)
Lung function data will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Lung function:
  FEV1, PEF, Oscillometry (daily)
Symptoms data (BCSS) will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  BCSS (daily)
Symptoms data (E-RS) will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  E-RS (daily)
Symptoms data (VAS-COPD) will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  VAS-COPD (daily)
Symptoms data (SGRQ) will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  SGRQ (fortnightly)
Symptoms data (CAT) will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  CAT (fortnightly)
Reliever use data will be plotted for each subject over the 12 weeks of the study to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Reliever use:
  Ventolin® use (daily)

SECONDARY OUTCOMES:
Inflammation data will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Inflammation:
  FeNO (daily) Blood eosinophils, CRP, and EDN (fortnightly) Sputum eosinophils and neutrophils (weekly)
Lung function data will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Lung function:
  FEV1, PEF, Oscillometry (daily)
Symptoms data (BCSS) will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  BCSS (daily)
Symptoms data (E-RS) will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  E-RS (daily)
Symptoms data (VAS-COPD) will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  VAS-COPD (daily)
Symptoms data (SGRQ) will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  SGRQ (fortnightly)
Symptoms data (CAT) will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  CAT (fortnightly)
Reliever use data will be plotted for a subject around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Reliever use:
  Ventolin® use (daily)

OTHER OUTCOMES:
Exploratory Biomarker data will be plotted for each subject over the 12 weeks of the study / around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Inflammation:
  Biomarkers from expectorate sputum samples (weekly) Biomarkers from nasal absorption samples (weekly) Plasma and serum exploratory biomarkers (fortnightly)
Exploratory Night time symptoms data will be plotted for each subject over the 12 weeks of the study / around a COPD worsening event to provide an understanding of the temporal dynamics of the data. | 12 weeks
  Symptoms:
  Night-time symptoms (passive monitoring, daily)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, Professor, Principal Investigator — Respiratory Department Churchill Hospital Old Road OX3 7LE
Locations (1):
- Research Site, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized indyvidual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment.:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. AZ will be accepting requests for IDP, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6930R00002&attachmentIdentifier=7135b354-0f60-4d34-9525-30cc4cea5f7d&fileName=d6930r00002-study-report-synopsis_for_redaction_Redactedv1.0A.pdf&versionIdentifier=